CLINICAL TRIAL: NCT06081842
Title: Strengthening Contraceptive Counseling Services, a Multi-country Study Trial
Brief Title: Strengthening Contraceptive Counseling Services: Research Protocol for a Multi-phase Complex Intervention in Pakistan and Nigeria
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: World Health Organization (Other)
Collaborators: Jinnah Sindh Medical University (Other); University of Ibadan (Other)
Responsible Party: Principal Investigator, Moazzam Ali, Medical officer / Epidemiologist, World Health Organization
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: WHO
Record Dates: First submitted 2023-09-18; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Contraception; Empowerment; Decision Making
Keywords: Family Planning, Counselling, choice
MeSH Terms: conditions — Empowerment

STUDY DESIGN:
Intervention Model Description: The research entails a complex multi-site, two-stage and 5-phase: STAGE 1 is formative and will comprise of a pre-formative (phase 1) and a formative (phase 2). While the STAGE 2 is experimental and will include intervention design (phase 3), experimental (phase 4), and reflective (phase 5).
Who Masked: Outcomes Assessor
Masking Description: Three-arm, single-blinded, parallel cluster randomized-controlled trial will compare routine care (arm 1) with the contraceptive counseling package (arm 2) and the same package combined with wider method availability (arm 3). Only data analysts will be masked to trial-arm allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1. Routine care (Active Comparator): Routine contraceptive counseling and routine method availability
  Interventions: Other: Contraceptive counseling strengthening intervention package
- Arm 2. Package of contraceptive counseling interventions (Experimental): The implementation package will be co-designed by providers and clients during the formative and research design phases
  Interventions: Other: Contraceptive counseling strengthening intervention package
- Arm 3. Expanded methods (Experimental): Routine care with the contraceptive counseling package combined with wider method availability as recommended by national policies.
  Interventions: Other: Contraceptive counseling strengthening intervention package

INTERVENTIONS:
Other: Contraceptive counseling strengthening intervention package — Development of contraceptive counseling strengthening intervention package that strengthens existing family planning services and is effective, safe, sustainable, scalable, and culturally appropriate.

SUMMARY:
High-quality contraceptive counseling can strengthen global efforts to reduce the unmet need for and suboptimal use of modern contraceptives. This study aims to identify a package of contraceptive counseling interventions for Pakistan and Nigeria designed to strengthen existing contraceptive services and determine its effectiveness in increasing clients' level of decision-making autonomy and meeting their contraceptive needs.

DETAILED DESCRIPTION:
The research will be a multi-intervention, three-arm, single-blinded, parallel, cluster RCT done in selected primary health centers (clusters) in Pakistan and in Nigeria. Centers will be randomly allocated to the three study arms in matched ratios (1:1:1) on the basis of the number of monthly family planning encounters, the number of available contraceptive types, the ratio of health workers per population in the clinic coverage zone, the location in urban or rural settings, and selected district-level variables that may have an influence on the study outcomes, including the unmet need for family planning, the level of literacy among women, and household income quartiles. Only data analysts will be masked to trial-arm allocation. Service providers skilled in family planning services will implement the clinical components of the contraceptive counseling package. The cluster RCT design is justified by the fact that some of the components of the intervention package to be identified in the intervention design phase will not be delivered directly to individual participants but only applied at the level of the health center, such as refresher training of service providers.

The two-part formative phase first uses participatory approaches to identify the perspectives of clients, including young people and providers, to ensure research contextualization and address each interest group's needs and priorities; clinical observations of client-provider encounters to document routine care form the second part. The design workshop of the third phase will result in the development of a package of contraceptive counseling interventions. In the fourth and experimental phase, a multi-intervention, three-arm, single-blinded, parallel cluster randomized-controlled trial will compare routine care (arm 1) with the contraceptive counseling package (arm 2) and the same package combined with wider method availability (arm 3). The fifth and reflective phase aims to analyze the package's cost-effectiveness and identify implementation barriers and enablers. The primary outcomes are clients' level of decision-making autonomy and met need for modern contraceptives.

ELIGIBILITY:
Inclusion Criteria:

1. Client comes to the family planning clinic with the intention to 1.a. use contraception for the first time in her life (new user), or 1.b. switch from a contraceptive method to another one (switching user), or 1.c. resume a method after not using any in the prior three months (lapse user), or 1.d. discontinue a modern method (discontinuing user);
2. Client is not coming for the resupply of a currently used method, such as pills or injectables;
3. Client has the intention to continue her follow-up at the health center during the duration of study follow-up;
4. Client does not participate in another study; and
5. Client provides informed consent.

Exclusion Criteria:

Not willing to participate in the complete duration of the trial

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 7920 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in clients' decision-making autonomy | Through study completion, an average of 1 year
  Person-Centered Contraceptive Counseling scale (PCCC). On a scale of 1-5, with score range between 4 to a maximum score of 20, with the highest possible score on a scale will be considered good.
Change in clients' met need for family planning | Through study completion, an average of 1 year
  Number of participants who want to avoid a pregnancy and are using a contraceptive method / all participants

SECONDARY OUTCOMES:
Change in modern contraceptive prevalence | 6 months and 12 months post enrollment
  Number of participants using a modern contraceptive / all participants

IPD SHARING:
Plan to Share IPD: Yes
(i) use of a controlled access approach, such as upon reasonable request from the World Health Organization; (ii) the trial will seek consent for sharing Individual Participant Data (IPD) from trial participants with adequate assurance that patient privacy and confidentiality will be maintained
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Supporting information will become available 6 months after data collection and will be available for at least 5 years
Access Criteria: Upon reasonable request from the World Health Organization

REFERENCES:
- [Derived] Tran NT, Ali M, Azmat SK, Seuc A, Olaolorun FM, Awan MA, Morhason-Bello I, Thom EM, Martin J, Abubakar HD, Uzma Q, Kiarie J. Strengthening contraceptive counselling services to empower clients and meet their needs: protocol for a two-stage, multiphase complex intervention in Pakistan and Nigeria. BMJ Open. 2024 Jun 5;14(6):e081967. doi: 10.1136/bmjopen-2023-081967. PMID 38839392